CLINICAL TRIAL: NCT06969287
Title: Mitigating Delirium With Fluvoxamine Treatment for Non-Cardiac Surgery (MD FluNCS)
Brief Title: Mitigating Delirium With Fluvoxamine Treatment for Non-Cardiac Surgery
Acronym: MD FluNCS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202411151; R21AG086855 (NIH)
Record Dates: First submitted 2025-04-30; First posted 2025-05-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Delirium; Surgery-Complications
Keywords: delirium; geriatric; surgery; fluvoxamine
MeSH Terms: conditions — Delirium | interventions — Fluvoxamine; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Oral Fluvoxamine 100 mg tablets (immediate release)
  Study drug (100mg Fluvoxamine tablet or placebo) will be administered at the following times:
  1. Day of surgery - Study drug to be taken morning of surgery and evening of surgery
  2. Post-operative day 1 - Study drug to be taken morning and evening
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants randomized using the randomization model in REDCAP. Study drug/placebo will be provided by an external pharmacy. Study drugs will be numbered and patients allocated to study drug using a randomisation model. Unblinding will only occur when the study finishes or if safety issues require.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluvoxamine (Experimental): 100 mg of fluvoxamine on the morning of surgery (POD 0), 100 mg on the evening of surgery (POD 0), 100 mg on the morning of POD 1, and 100 mg on the evening of POD 1. All administered as PO capsules.
  Interventions: Drug: Fluvoxamine
- Placebo (Placebo Comparator): Placebo capsule on the morning of surgery (POD 0), Placebo capsule on the evening of surgery (POD 0), Placebo capsule on the morning of POD 1, and Placebo capsule on the evening of POD 1. All administered PO.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine — 100mg Fluvoxamine Capsule
  1. Day of surgery - Study drug to be taken morning of surgery and evening of surgery
  2. Post-operative day 1 - Study drug to be taken morning and evening
  Other Names: Oral Fluvoxamine 100 mg capsules (immediate release)
  Arms: Fluvoxamine
Drug: Placebo — Placebo Capsule
  1. Day of surgery - Study drug to be taken morning of surgery and evening of surgery
  2. Post-operative day 1 - Study drug to be taken morning and evening
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The investigation will establish biological plausibility and infrastructure required for a multisite clinical trial evaluating the re-purposing of fluvoxamine to mitigate postoperative delirium risk in geriatric patients undergoing non-cardiac non-intracranial surgery.

DETAILED DESCRIPTION:
Delirium is a disturbance in attention, cognition, and consciousness, an acute physiological consequence of medical events, such as hospital admission, surgery, sepsis, and pharmacological intervention. There are currently no standard pharmacologic interventions to prevent delirium in any setting. The investigation will lay the groundwork for a larger-scale Phase 3 trial geared toward advancing long-term goal of improving public health and quality of life for those at risk of postoperative delirium and related sequelae.

The study assumes that neuroinflammation is a key contributor to the pathogenesis of postoperative delirium, a matter of conjecture. The investigators will directly test systemic inflammation as a proxy for neuroinflammation. The investigation will test whether fluvoxamine may be associated with reduced systemic inflammation, markers of neural dysfunction, and delirium severity.

This potential therapeutic approach has potential generalizability to different clinical settings and already proved useful for COVID-19. The investigators combine the need to develop a collaborative clinical trials platform across diverse healthcare settings with key mechanistic studies that will advance our understanding of the pathogenesis of delirium. These studies will leverage high-density EEG recordings and state-of-the-art plasma biomarker collection, providing key data on the biological plausibility for a fluvoxamine effect.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* elective non-cardiac or non-intracranial surgery requiring at least a 2-day hospital length of stay

Exclusion Criteria:

* Received investigational drug within the last 7 weeks
* lack of capacity to provide informed consent
* prior known intolerance or allergy to SSRIs or fluvoxamine
* planned postoperative ventilation
* drug or alcohol dependence
* preoperative use of non-NSAID medications with drug-drug interactions of Class X (Avoid Combination) or D (Consider Therapy Modification)
* risk of serotonin syndrome (St John's Wort, SSRIs, or TCA)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Average Monthly participant enrollment rate | 12- months, duration of the study
  Feasibility assessed as number of eligible participants enrolled per month by an audit of the study screening and recruitment logs.

SECONDARY OUTCOMES:
Average Monthly screen failure rate | 12- months, duration of the study
  Feasibility assessed as number of screening failures per month by an audit of the study screening and recruitment logs.
Average Monthly rate of withdrawal | 12- months, duration of the study
  Feasibility assessed as number of withdrawals per month by an audit of the study screening and recruitment logs.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be released in manuscript form. Outcome data will be uploaded to the OpenNeuro on a rolling basis.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within three years of study completion
Access Criteria: Data use agreements may be required.